CLINICAL TRIAL: NCT03123471
Title: A Phase 3, Multi-Center, Randomized, Placebo-Controlled, Double-Blind, Study of the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Moderate to Severe Plaque Psoriasis of the Scalp
Brief Title: A Study of the Efficacy and Safety of Apremilast (CC-10004) in Subjects With Moderate to Severe Plaque Psoriasis of the Scalp
Acronym: STYLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-SPSO-001; U1111-1194-1248 (Registry Identifier: WHO)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Scalp; Double-Blind; Efficacy; Safety; CC-10004; Apremilast; Otezla; Itch; Head
MeSH Terms: conditions — Psoriasis; Pruritus | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apremilast 30 mg BID (Experimental): Apremilast 30 mg tablets orally twice daily (BID) during Weeks 0 to 32
  Interventions: Drug: Apremilast; Other: Placebo
- Placebo (Placebo Comparator): Placebo tablets BID during weeks 0 to 16; at week 16, placebo participants were switched to apremilast 30 mg tablets BID for 16 weeks (from Week 16 to Week 32)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg tablets BID from weeks 0 to 32.
  Other Names: CC-10004
  Arms: Apremilast 30 mg BID
Other: Placebo — Placebo tablets twice daily (BID) for 16 weeks; placebo participants were switched to apremilast 30 mg at week 16.

SUMMARY:
This is a Phase 3, multicenter, randomized, placebo-controlled, double-blind study of the efficacy and safety of apremilast (CC-10004) in subjects with moderate to severe plaque psoriasis of the scalp.

Approximately 300 subjects with moderate to severe plaque psoriasis of the scalp will be randomized 2:1 to receive either apremilast 30 mg twice daily (BID) or placebo for the first 16 weeks.

DETAILED DESCRIPTION:
The study will consist of four phases:

* Screening Phase - up to 35 days
* Double-blind Placebo-controlled Phase- Weeks 0 to 16 Subjects will receive treatment with one of the following:

  * apremilast 30 mg tablets orally BID or
  * placebo tablets (identical in appearance to apremilast 30 mg tablets) orally BID
* Apremilast Extension Phase - Weeks 16 to 32

  * All subjects who had received placebo during the placebo-controlled phase will be switched to apremilast 30 mg BID (or continue with) apremilast. At Week 16, all subjects will maintain this dosing through Week 32.
* Observational Follow-up Phase

  * Four-week Post-Treatment Observational Follow-up Phase for all subjects who complete the study or discontinue from the study early.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Males or females, ≥ 18 years of age at the time of signing the informed consent document
* Be willing and able to adhere to the study visit schedule and other protocol requirements.
* Have a diagnosis of moderate to severe plaque psoriasis of the scalp at screening and baseline
* Must be a candidate for phototherapy and/or systemic therapy for either body or scalp psoriasis lesions.
* Have moderate to severe plaque psoriasis at screening and baseline
* Must be in good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), clinical laboratories, and urinalysis
* Must meet laboratory criteria
* Females of childbearing potential (FCBP)* must have a negative pregnancy test at screening and baseline. While on investigational product (IP) and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible - must use one of the approved contraceptive** options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

*A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

** The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Other than psoriasis, history of any clinically significant uncontrolled disease.

Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.

* Pregnant or breast feeding
* Hepatitis B surface antigen positive at screening
* Anti-hepatitis C antibody positive at screening
* Active tuberculosis (TB) or a history of incompletely treated TB
* Clinically significant abnormality on 12-lead electrocardiogram (ECG) at screening
* History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease)
* Active substance abuse or a history of substance abuse within 6 months prior to signing the informed consent form.
* Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of signing the informed consent form.
* Malignancy or history of malignancy, except for treated (i.e., cured) basal cell or squamous cell in situ skin carcinomas or treated (i.e., cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within 5 years of signing the informed consent.
* Prior history of suicide attempt at any time in the subject's life time prior to signing the informed consent and randomization, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
* Psoriasis flare/rebound within 4 weeks of signing the informed consent form or between the screening and baseline visits.
* Topical therapy within 2 weeks prior to randomization; Conventional systemic therapy for psoriasis within 4 weeks prior to randomization; Intralesional corticosteroids on the scalp within 2 weeks prior to randomization; Phototherapy treatment of body or scalp psoriasi lesions within 4 weeks prior to randomization; Biologic therapy between 12 weeks to 24 weeks prior to randomization
* Use of any investigational drug beginning 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer)
* Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources
* Prior treatment with apremilast
* History of allergy or hypersensitivity to any components of the Investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- United States (31):
  - Northwest Arkansas Clinical Trials Center, PLLC / Hull Dermatology, Rogers, Arkansas
  - Tien Q. Nguyen MD Inc, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - San Luis Dermatology and Laser Clinic, San Luis Obispo, California
  - University of Connecticut, Farmington, Connecticut
  - Florida Academic Centers Research and Education, Coral Gables, Florida
  - International Dermatology Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Dermatologic Surgery Specialists, P.C., Macon, Georgia
  - MedaPhase INC, Newnan, Georgia
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Lawrence Green, MD, LLC, Rockville, Maryland
  - Central Dermatology, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Icahn School of Medicine at Mount Sinai Medical Center, New York, New York
  - Sadick Research Group, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Wright State Physicians, Fairborn, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Austin Dermatology Associates, Austin, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Clinical Research Inc, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (13):
  - Kirk Barber Research, Calgary, Alberta
  - Institute for Skin Advancement, Calgary, Alberta
  - Chih-Ho Hong Medical, Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research, Markham, Ontario
  - North Bay Dermatology Center, North Bay, Ontario
  - Skin Center for Dermatology, Peterborough, Ontario
  - Centre For Dermatology and Cosmetic Surgery, Richmond Hill, Ontario
  - The Toronto Dermatology Centre, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain CRDQ, Québec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Wang Y, Coyne K, Sofen H, Santanello N, Currie B, Zhang Z, Nograles K. Qualitative analysis and reproducibility assessment of the Scalp Itch Numeric Rating Scale among patients with moderate to severe plaque psoriasis of the scalp. J Dermatolog Treat. 2019 Dec;30(8):775-783. doi: 10.1080/09546634.2019.1577546. Epub 2019 Mar 5. PMID 30747550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 303 participants were randomized to study treatment at 41 sites in the United States and Canada.
Pre-assignment Details: Participants were randomly assigned in a 2:1 ratio to receive either apremilast or placebo. Randomization was stratified by baseline Scalp Physician Global Assessment (ScPGA) score (moderate [3], severe [4]) to ensure balance between treatment arms with respect to baseline severity of scalp psoriasis.
Groups:
- Placebo/Apremilast: Participants received identically matching placebo capsules twice daily (BID) during the placebo-controlled phase. At week 16, participants were switched to apremilast 30 mg capsules BID during the apremilast extension treatment phase and received apremilast from week 16 to week 32.
- Apremilast: Participants received apremilast 30 mg capsules BID during the 16-week placebo-controlled phase and continued to receive apremilast 30 mg BID capsules during the apremilast extension phase from week 16 to week 32.
Period: Placebo-controlled Phase
Arm/Group | Placebo/Apremilast | Apremilast
Started | 102 | 201
Received at Least 1 Dose of Study Drug | 102 | 200
Completed | 84 | 168
Not Completed | 18 | 33
Not completed — Adverse Event | 3 | 8
Not completed — Lack of Efficacy | 3 | 4
Not completed — Withdrawal by Subject | 6 | 16
Not completed — Non-compliance with Study Drug | 3 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Deviation | 2 | 1
Not completed — Miscellaneous | 0 | 1
Period: Apremilast Extension Phase
Arm/Group | Placebo/Apremilast | Apremilast
Started | 84 | 165 (3 participants completed the first phase; did not enter in extension phase)
Received at Least 1 Dose of Study Drug | 84 | 163
Completed | 76 | 140
Not Completed | 8 | 25
Not completed — Lost to Follow-up | 2 | 5
Not completed — Adverse Event | 1 | 5
Not completed — Lack of Efficacy | 2 | 8
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Apremilast | Apremilast | Total
Number analyzed (Participants) | 102 | 201 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (15.15) | 47.0 (15.02) | 46.9 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 76 | 116
  Male | 62 | 125 | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 27 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 75 | 154 | 229
  Black or African American | 7 | 12 | 19
  Other | 4 | 4 | 8
  Unknown or Not Reported | 0 | 2 | 2
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: Years] | 14.75 (11.262) | 15.67 (12.405) | 15.36 (12.022)
Scalp Physician Global Assessment (ScPGA) Score [Count of Participants; unit: Participants] — The ScPGA is a measurement of overall scalp involvement by the investigator at the time of evaluation. The ScPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling, and plaque elevation.
  Participants
    0 (Clear) | 0 | 0 | 0
    1 (Almost Clear) | 0 | 0 | 0
    2 (Mild) | 0 | 0 | 0
    3 (Moderate) | 78 | 155 | 233
    4 (Severe) | 24 | 46 | 70
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was based on the last weight and height measurement taken prior to the randomization date.
  kg/m^2 | 31.66 (7.175) | 30.66 (7.100) | 31.00 (7.129)
Whole Body Itch Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: Units on a Scale] — The Whole-Body Itch NRS scale is a 11-point scale to assess whole body itch. The scale ranges from 0-10, where "0" represents no itch, and "10" represents the worst imaginable itch, and a 4-point change from baseline was shown to be optimal for demonstrating a level of clinically meaningful improvement in itch severity.
  Units on a Scale | 7.2 (1.99) | 7.2 (2.25) | 7.2 (2.16)
Scalp Itch NRS Score [Mean (Standard Deviation); unit: Units on a Scale] — The scalp itch NRS is a 11-point scale to assess scalp itch. The scale ranges from 0-10, where "0" represents no itch, and "10" represents the worst imaginable itch
  Units on a Scale | 6.7 (2.41) | 6.6 (2.49) | 6.7 (2.46)
Dermatological Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: Units on a Scale] — DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of various skin diseases. The instrument contains ten items assessed on a QOL scale dealing with the participant's skin. The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
  Units on a Scale | 12.6 (7.20) | 12.6 (7.03) | 12.6 (7.07)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Scalp Physician Global Assessment (ScPGA) Score of Clear (0) or Almost Clear (1) With at Least a 2-Point Reduction From Baseline
Description: The ScPGA is a measurement of overall scalp involvement by the investigator at the time of evaluation. The ScPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the 3 primary signs of the disease: erythema, scaling, and plaque elevation. When making the assessment of overall scalp severity, the investigator factored in areas that had already been cleared (ie, had scores of 0), not limited to the evaluation of remaining lesions for severity; consequently, the severity of each sign was averaged across all areas of involvement, including cleared lesions.
Time Frame: Baseline to Week 16
Population: The intent to treat (ITT) population included participants who were randomized. Missing values were imputed using the multiple imputation (MI) method.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 102 | 201
Percentage of Participants | 13.7 [6.6 to 20.8] | 43.3 [36.2 to 50.5]
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Apremilast; The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and the 2-sided 95% confidence interval using a normal approximation to the weighted average were calculated; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 29.6, 95% CI 2-sided [19.5 to 39.7]

2. Secondary Outcome: Percentage of Participants With ≥ 4-Point Reduction (Improvement) From Baseline in the Whole Body Itch Numeric Rating Score at Week 16
Description: The Whole Body Itch NRS scale is an 11-point scale to assess whole body itch. The scale ranges from 0-10, where "0" represents no itch, and "10" represents the worst imaginable itch, and a 4-point change from baseline was shown to be optimal for demonstrating a level of clinically meaningful improvement in itch severity. NRS response was defined as a ≥ 4-point reduction (improvement) from baseline.
Time Frame: Baseline to Week 16
Population: Participants in the ITT population who had a baseline Body Itch NRS Score ≥4. Missing values were imputed using the multiple imputation method.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 94 | 185
Percentage of Participants | 22.5 [13.7 to 31.3] | 45.5 [38.1 to 52.9]
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Apremilast; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 23.0, 95% CI 2-sided [11.5 to 34.6]

3. Secondary Outcome: Percentage of Participants With ≥ 4-Point Reduction (Improvement) From Baseline in the Scalp Itch Numeric Rating Score (NRS) at Week 16
Description: The scalp itch NRS is a 11-point scale to assess scalp itch. The scale ranges from 0-10, where "0" represents no itch, and "10" represents the worst imaginable itch.
Time Frame: Baseline to Week 16
Population: Includes participants in the ITT population had baseline scalp itch NRS Score ≥ 4. Missing values were imputed using the multiple imputation method.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 90 | 175
Percentage of Participants | 21.1 [11.8 to 30.3] | 47.1 [39.5 to 54.7]
Statistical Analysis 1: Comparison: Apremilast; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 26.2, 95% CI 2-sided [13.9 to 38.5]

4. Secondary Outcome: Percentage of Participants With ≥ 4-Point Reduction (Improvement) From Baseline in the Whole Body Itch NRS Score by Visit in the Placebo-Controlled Phase
Description: The Whole Body Itch NRS scale is a 11-point scale to assess whole body itch. The scale ranges from 0-10, where "0" represents no itch, and "10" represents the worst imaginable itch, and a 4-point change from baseline was shown to be optimal for demonstrating a level of clinically meaningful improvement in itch severity.
Time Frame: Baseline to Weeks 2, 4, 6, 8 and 12
Population: Participants in the ITT population with a baseline whole body itch NRS Score ≥ 4. Missing values were imputed using the multiple imputation method.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 94 | 185
Percentage of Participants
  Week 2 | 3.5 [-0.4 to 7.4] | 20.5 [14.6 to 26.4]
  Week 4 | 10.1 [3.9 to 16.3] | 32.3 [25.4 to 39.1]
  Week 8 | 19.7 [11.4 to 27.9] | 39.8 [32.6 to 47.1]
  Week 12 | 26.3 [17.0 to 35.7] | 47.0 [39.6 to 54.3]
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Apremilast; Week 2; The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and the 2-sided 95% confidence interval using a normal approximation to the weighted average were calculated; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 17.0, 95% CI 2-sided [9.8 to 24.2]
Statistical Analysis 2: Comparison: Placebo/Apremilast vs Apremilast; Week 4. The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and the 2-sided 95% confidence interval using a normal approximation to the weighted average were calculated; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 22.1, 95% CI 2-sided [12.9 to 31.4]
Statistical Analysis 3: Comparison: Placebo/Apremilast vs Apremilast; Week 8; The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and the 2-sided 95% confidence interval using a normal approximation to the weighted average were calculated; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 20.1, 95% CI 2-sided [9.1 to 31.0]
Statistical Analysis 4: Comparison: Placebo/Apremilast vs Apremilast; Week 12; The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and SE using a normal approximation to the weighted average were calculated; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 20.6, 95% CI 2-sided [8.7 to 32.4]

5. Secondary Outcome: Percentage of Participants With ≥ 4-Point Reduction (Improvement) From Baseline in the Scalp Itch NRS Score by Visit in the Placebo-Controlled Phase
Description: as for outcome 3
Time Frame: Baseline to Weeks 2, 4, 8 and 12
Population: The intent to treat population included participants who were randomized; analysis includes participants with a baseline scalp itch NRS Score ≥4. Missing values were imputed using the multiple imputation method.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 90 | 175
Percentage of Participants
  Week 2 | 11.5 [4.8 to 18.2] | 26.1 [19.5 to 32.7]
  Week 4 | 16.5 [8.7 to 24.4] | 37.8 [30.5 to 45.0]
  Week 8 | 23.7 [14.6 to 32.9] | 45.6 [38.1 to 53.2]
  Week 12 | 19.6 [10.6 to 28.5] | 46.5 [38.9 to 54.1]
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Apremilast; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 14.6, 95% CI 2-sided [5.1 to 24.1]
Statistical Analysis 2: Comparison: Placebo/Apremilast vs Apremilast; Week 4; The adjusted difference in response rates using the weighted average of the treatment differences across the strata with the CMH weights and the 2-sided 95% confidence interval using a normal approximation to the weighted average were calculated; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 21.3, 95% CI 2-sided [10.6 to 31.9]
Statistical Analysis 3: Comparison: Placebo/Apremilast vs Apremilast; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 22.0, 95% CI 2-sided [10.2 to 33.9]
Statistical Analysis 4: Comparison: Placebo/Apremilast vs Apremilast; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Analysis used CMH; adjusted by stratification factor of baseline ScPGA score moderate (3) or severe (4); Difference in Response = 27.0, 95% CI 2-sided [15.1 to 38.9]

6. Secondary Outcome: Change From Baseline in Dermatological Life Quality Index (DLQI) Total Score at Week 16
Description: DLQI is questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the subject is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score was derived by summing all item scores, and has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline to Week 16
Population: The intent to treat population included participants who were randomized. Missing values were imputed using the multiple imputation method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 102 | 201
Units on a Scale | -3.8 (0.56) | -6.7 (0.41)
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Apremilast; Test type: Superiority; p < 0.0001, ANCOVA; Treatment and stratification factor (Baseline ScPGA moderate or severe) as independent variables and baseline value as a covariate variable; Difference in LS Mean = -2.9, 95% CI 2-sided [-4.17 to -1.73]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Placebo-Controlled Phase
Description: A TEAE is an AE with a start date on or after the date of the first dose of study drug and no later than 28 days after the last dose of study drug. A serious AE (SAE) is any untoward AE that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize or may require intervention to prevent one of the outcomes above. The severity of AEs was assessed based on the following scale: Mild = asymptomatic or mild symptoms, clinical or diagnostic observations only; Moderate = symptoms cause moderate discomfort; Severe = could be non-serious or serious) = symptoms causing severe pain discomfort.
Time Frame: Week 0 to Week 16; mean duration of exposure was 14.5 weeks and 14.6 weeks for participants randomized to placebo and apremilast respectively.
Population: Safety population includes participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast | Placebo/Apremilast
Number analyzed (Participants) | 200 | 102
Participants
  Any TEAE | 135 | 52
  Any Drug-related TEAE | 99 | 22
  Any Severe TEAE | 5 | 2
  Any Serious TEAE | 2 | 1
  Any TEAE Leading to Drug Interruption | 9 | 4
  Any TEAE Leading to Drug Withdrawal | 11 | 3

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Apremilast-Extension Phase
Description: as for outcome 7
Time Frame: Weeks 16 to Week 32; the mean treatment duration was 14.6 weeks and 15.3 weeks in the APR 30/APR 30 BID and placebo/APR 30 BID arms, respectively
Population: Safety population includes participants who received at least 1 dose of study drug. Participants who entered into the apremilast extension phase and were treated.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast: Participants randomized to apremilast 30 mg capsules BID during the placebo-controlled phase and continued to receive apremilast 30 mg BID capsules from week 16 to week 32
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 84 | 163
Participants
  Any TEAE | 35 | 66
  Any Drug-related TEAE | 17 | 17
  Any Severe TEAE | 2 | 4
  Any Serious TEAE | 1 | 5
  Any TEAE Leading to Drug Interruption | 2 | 4
  Any TEAE Leading to Drug Withdrawal | 1 | 4
  Deaths | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Apremilast-Exposure Period
Description: The apremilast-exposure period started on the date of the first dose of apremilast (Week 0 for participants originally randomized to apremilast or Week 16 for participants originally randomized to placebo) to the last dose of apremilast. A TEAE is an AE with a start date on or after the date of the first dose of study drug and no later than 28 days after the last dose of study drug. A serious AE (SAE) is any untoward AE that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize or may require intervention to prevent one of the outcomes above. The severity of AEs was assessed based on the following scale: Mild = asymptomatic or mild symptoms, clinical or diagnostic observations only; Moderate = symptoms cause moderate discomfort; Severe = could be non-serious or serious) = symptoms causing severe pain discomfort.
Time Frame: Week 0 to 32;
Population: The apremilast participants as treated population, which includes all participants who were randomized to (at Week 0) or treated with (at Week 16) apremilast 30 mg BID, and received at least one dose of apremilast after randomization or Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Apremilast | Apremilast
Number analyzed (Participants) | 84 | 200
Participants
  Any TEAE | 35 | 144
  Any Drug-related TEAE | 17 | 103
  Any Severe TEAE | 2 | 8
  Any Serious TEAE | 1 | 6
  Any Serious TEAE Drug Related TEAE | 0 | 3
  Any TEAE Leading to Drug Interruption | 2 | 13
  Any TEAE Leading to Drug Withdrawal | 1 | 15
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of randomization to 28 days after the last dose of study drug. AEs are reported for the placebo-controlled phase from Week 0 to Week 16 and for the apremilast extension phase from Week 16 to Week 32;
Description: AEs are reported for the Apremilast Exposure Period from Week 0 to Week 32; the mean treatment duration to apremilast was 23.2 weeks.
Groups:
- Placebo (Weeks 0-16): Participants received identically matching placebo capsules twice daily during the 16-week placebo-controlled phase.
- Apremilast 30 mg (Weeks 0-16): Participants received apremilast 30 mg capsules BID during the 16-week placebo-controlled phase.
- Placebo/Apremilast (APR Extension Phase Weeks 16-32): Participants initially randomized to placebo capsules BID during the placebo controlled phase were switched to apremilast 30 mg capsules BID at week 16 and continued apremilast up to Week 32.
- Apremilast /Apremilast (APR Exposure Period, Weeks 0-32): Participants received apremilast 30 mg capsules BID during the placebo-controlled phase and continued to receive apremilast 30 mg BID capsules from weeks 16 to week 32.
- Apremilast Total (APR Exposure Period, Weeks 0-32): Participants who started apremilast 30 mg BID at any time during the study (Week 0 for participants originally randomized to apremilast or at week 16 for participants originally randomized to placebo.
Arm/Group | Placebo (Weeks 0-16) | Apremilast 30 mg (Weeks 0-16) | Placebo/Apremilast (APR Extension Phase Weeks 16-32) | Apremilast /Apremilast (APR Exposure Period, Weeks 0-32) | Apremilast Total (APR Exposure Period, Weeks 0-32)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/200 | 0/84 | 0/200 | 0/284
Serious Adverse Events (participants affected / at risk) | 1/102 | 2/200 | 1/84 | 6/200 | 7/284
Other Adverse Events (participants affected / at risk) | 23/102 | 95/200 | 19/84 | 101/200 | 120/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=102) | Apremilast 30 mg (Weeks 0-16) (N=200) | Placebo/Apremilast (APR Extension Phase Weeks 16-32) (N=84) | Apremilast /Apremilast (APR Exposure Period, Weeks 0-32) (N=200) | Apremilast Total (APR Exposure Period, Weeks 0-32) (N=284)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=102) | Apremilast 30 mg (Weeks 0-16) (N=200) | Placebo/Apremilast (APR Extension Phase Weeks 16-32) (N=84) | Apremilast /Apremilast (APR Exposure Period, Weeks 0-32) (N=200) | Apremilast Total (APR Exposure Period, Weeks 0-32) (N=284)
Diarrhoea (Gastrointestinal disorders) | 11 | 61 | 14 | 62 | 76
Nausea (Gastrointestinal disorders) | 6 | 43 | 8 | 47 | 55
Vomiting (Gastrointestinal disorders) | 2 | 11 | 2 | 13 | 15
Fatigue (General disorders) | 4 | 9 | 2 | 12 | 14
Influenza (Infections and infestations) | 2 | 8 | 2 | 10 | 12
Headache (Nervous system disorders) | 5 | 24 | 3 | 25 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT03123471/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03123471/SAP_001.pdf